CLINICAL TRIAL: NCT02284906
Title: A Blinded Long-term Extension Study to Evaluate the Safety and Efficacy of Pioglitazone (AD-4833 Sustained Release 0.8 mg Daily) to Slow the Progression of Cognitive Decline in Subjects Who Have Completed the AD-4833/TOMM40_301 Study With Diagnosis of Mild Cognitive Impairment Due to Alzheimer Disease
Brief Title: AD-4833/TOMM40_303 Extension Study of the Safety and Efficacy of Pioglitazone to Slow Cognitive Decline in Participants With Mild Cognitive Impairment Due to Alzheimer Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy of the drug; no safety concern
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AD-4833/TOMM40_303; U1111-1154-9637 (Registry Identifier: WHO); 2013-004984-30 (EudraCT Number)
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Mild Cognitive Impairment Due to Alzheimer's Disease
Keywords: Drug therapy
MeSH Terms: interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Pioglitazone 0.8 mg (Experimental): Pioglitazone 0.8 mg, tablets, orally, once, daily, for minimum of 2 years.
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator): Pioglitazone placebo-matching tablets, orally, once, daily, for minimum of 2 years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone tablets
  Other Names: AD-4833
  Arms: Pioglitazone 0.8 mg
Drug: Placebo — Pioglitazone placebo-matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of pioglitazone at 24 months compared with placebo on cognitive decline in high-risk participants who have completed the AD-4833/TOMM40_301 study [NCT01931566] with an adjudicated diagnosis of mild cognitive impairment (MCI) due to Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
The drug being tested in this study is called pioglitazone. This study is designed to further evaluate the safety and effectiveness of pioglitazone on cognitive function in participants who have completed the AD-4833/TOMM40_301. This study will look at the effectiveness of pioglitazone on cognitive decline in high-risk participants who have completed the AD-4833/TOMM40_301 study with a diagnosis of mild cognitive impairment (MCI) due to Alzheimer's Disease (AD).

The study enrolled 40 participants, but is dependent on how many decide to continue treatment in an extension phase after completing the main (301) study. Participants will continue to receive the same study medication they received during the pivotal AD-4833/TOMM40_301 study, either:

* Pioglitazone 0.8 mg tablets or
* Placebo (this is a tablet that looks like the study drug but has no active ingredient).

All participants will be asked to take one tablet at the same time each day throughout the study.

This multi-centre trial, like its precedent pivotal trial, will be conducted worldwide. The overall time to participate in this study is minimum 2 years and a maximum of 7 years depending on when participants roll over from the 301 study. Participants will make approximately 2 visits per year to the clinic, and will be contacted by telephone 3 months after each treatment visit for a follow-up assessment, and 2 weeks after the final visit.

ELIGIBILITY:
Inclusion Criteria:

1. Completed the pivotal AD-4833/TOMM40_301 study with an adjudicated diagnosis of mild cognitive impairment (MCI) due to Alzheimer's Disease (AD) without ongoing serious adverse events (SAEs) from AD-4833/TOMM40_301.
2. Is male or female and is at least 65 years of age at the time of the Baseline Visit.
3. In the opinion of the investigator, is capable of understanding and complying with the protocol requirements.
4. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
5. Must be living independently or in nonmedical residential care.
6. Has a project partner able to separately consent on his/her own behalf and take part in the study (with the intent to do so as long as the participant is enrolled), providing information on the cognitive, functional, and behavioral status of the participant and assisting with observation of adverse events (AEs) and monitoring of study medication, if needed. Project partners participating in the pivotal AD-4833/TOMM40_301 study are encouraged to participate in this extension study in this capacity.

Exclusion Criteria:

1. Completed the pivotal AD-4833/TOMM40_301 study with an adjudicated diagnosis of AD dementia.
2. Has a current diagnosis of significant psychiatric illness, per Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (including but not limited to major depressive disorder, anxiety disorders) and is in an acute phase/episode, or the participant has a current diagnosis or history of schizophrenia or bipolar disorder.
3. Has a glycosylated hemoglobin (HbA1c) >8% at the extension study Baseline Visit or requires treatment with insulin, triple oral antidiabetic therapy or a peroxisome proliferator-activated receptor gamma (PPAR-γ) agonist.
4. Has a clinically significant unstable illness, for example, hepatic impairment or renal insufficiency, or cardiovascular, pulmonary, gastrointestinal (including s/p gastric bypass surgery), endocrine, neurological, rheumatologic, immunologic, infectious, skin and subcutaneous tissue disorders, or metabolic disturbance.
5. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (eg, spouse, pivotal, child, sibling) or may consent under duress.
6. Is required to take excluded medications.
7. Has a history of hypersensitivity or allergies to pioglitazone or related compounds.
8. Had any of the following values at the extension study Baseline Visit:

   1. A serum total bilirubin value >15 x upper limit of normal (ULN).
   2. A serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value >2 x ULN.
   3. Unexplained microscopic/macroscopic hematuria on 2 repeat examinations within 2 weeks.
9. Has a disease or takes medication that, in the opinion of the investigator, could interfere with the assessments of safety, tolerability, or efficacy, or prevent the participant from adequately participating in the study or continue for the anticipated duration of the study.
10. Has received any investigational compound, with the exception of treatment during the AD-4833/TOMM40_301 study, within 30 days prior to Baseline or 5 half-lives prior to Baseline or is currently participating in another study that entails the administration of an investigational or marketed drug, supplement, or intervention including, but not limited to diet, exercise, lifestyle, or invasive procedure.
11. Has any cancer that has been in remission for less than 2 years from the extension study Baseline Visit. Participants with basal cell or stage I squamous cell carcinoma of the skin will be eligible. Participants with current diagnosis of bladder cancer are not eligible irrespective of the remission status.
12. Has a current diagnosis of macular edema, degeneration or any maculopathy.
13. Has a history or current diagnosis of congestive heart failure (CHF), New York Heart Association class III-IV.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02-12 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (43):
- United States (28):
  - Phoenix, Arizona
  - Sun City, Arizona
  - San Diego, California
  - Delray Beach, Florida
  - Fort Myers, Florida
  - Lake Worth, Florida
  - Melbourne, Florida
  - Merritt Island, Florida
  - Port Orange, Florida
  - St. Petersburg, Florida
  - Weston, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Chicago, Illinois
  - Elk Grove, Illinois
  - Elk Grove Village, Illinois
  - Iowa City, Iowa
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Marlton, New Jersey
  - New York, New York
  - Concord, North Carolina
  - Durham, North Carolina
  - Akron, Ohio
  - Charleston, South Carolina
  - Houston, Texas
  - Salt Lake City, Utah
  - Middleton, Wisconsin
- Australia (4):
  - North Ryde, New South Wales
  - Southport, Queensland
  - Heidelberg West, Victoria
  - Nedlands, Western Australia
- Basel, Switzerland
- United Kingdom (10):
  - Bristol, Avon
  - Exeter, Devon
  - Plymouth, Devon
  - Hammersmith, Greater London
  - London, Greater London
  - Manchester, Greater Manchester
  - Blackpool, Lancashire
  - Isleworth, Middlesex
  - Glasgow, Strathclyde
  - Perth, Tayside Region

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 3 investigative sites in Australia, United Kingdom and United States from 12 Feb 2015 to 08 May 2018.
Pre-assignment Details: Participants with who have completed the pivotal AD-4833/TOMM40_301 (NCT01931566) study with an adjudicated diagnosis of mild cognitive impairment (MCI) due to Alzheimer's Disease (AD) were enrolled to pioglitazone (0.8 mg sustained release tablet) or placebo.
Groups:
- Low Risk Placebo: Pioglitazone placebo-matching tablets, orally, once daily, for 10 months to participants assigned to low risk group for developing MCI- AD within the next five years in previous study (AD-4833/TOMM40_301).
- High Risk Placebo: Pioglitazone placebo-matching tablets, orally, once daily, for minimum of 3 years to participants assigned to high risk group for developing MCI- AD within the next five years in previous study (AD-4833/TOMM40_301).
- High Risk Pioglitazone: Pioglitazone 0.8 mg tablets, orally, once daily for 3 years to participants assigned to high risk group for developing MCI- AD within the next five years in previous study (AD-4833/TOMM40_301).
Period: Overall Study
Arm/Group | Low Risk Placebo | High Risk Placebo | High Risk Pioglitazone
Started | 3 | 18 | 19
Completed | 0 | 0 | 0
Not Completed | 3 | 18 | 19
Not completed — Pretreatment Event/Adverse Event | 0 | 1 | 0
Not completed — Major Protocol Deviation | 0 | 1 | 0
Not completed — Voluntary Withdrawal | 2 | 4 | 5
Not completed — Study Termination | 0 | 11 | 14
Not completed — Reason not Specified | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of blinded study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Risk Placebo | High Risk Placebo | High Risk Pioglitazone | Total
Number analyzed (Participants) | 3 | 18 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.7 (4.73) | 78.9 (3.98) | 78.1 (4.42) | 78.2 (4.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 10 | 16
  Male | 2 | 13 | 9 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 2 | 17 | 18 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 0 | 0 | 1 | 1
  White | 3 | 18 | 18 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic/Latino Caucasian | 2 | 17 | 17 | 36
  Hispanic/Latino and/or non-Caucasian | 1 | 1 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 11 | 15 | 28
  United Kingdom | 1 | 2 | 2 | 5
  Australia | 0 | 5 | 2 | 7
Height [Mean (Standard Deviation); unit: cm] | 169.7 (4.16) | 168.7 (10.85) | 166.8 (11.73) | 167.9 (10.81)
Weight [Mean (Standard Deviation); unit: kg] | 78.20 (6.053) | 76.00 (13.719) | 72.11 (15.685) | 74.32 (14.224)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI=Weight/Height^2. Both weight and height measurements were from extension study baseline, which was conducted at the End of Study visit for the pivotal AD-4833/TOMM40_301 study.
  kg/m^2 | 27.27 (3.412) | 26.49 (2.769) | 25.68 (3.653) | 26.16 (3.218)
Smoking Classification [Count of Participants; unit: Participants]
  Participant Has Never Smoked | 2 | 7 | 9 | 18
  Participant is an Ex-smoker | 1 | 11 | 10 | 22
Alcohol Classification [Count of Participants; unit: Participants]
  Participant Has Never Drunk | 1 | 3 | 3 | 7
  Participant is a Current Drinker | 2 | 15 | 15 | 32
  Participant is an Ex-drinker | 0 | 0 | 1 | 1
Years of Education [Mean (Standard Deviation); unit: years] | 15.0 (3.61) | 14.8 (3.59) | 14.9 (3.67) | 14.9 (3.54)
Years Lived in Country/Region for 10 Years or More [Count of Participants; unit: Participants] | 3 | 18 | 19 | 40
Primary Language [Count of Participants; unit: Participants]
  English | 2 | 16 | 19 | 37
  Other | 1 | 2 | 0 | 3
Ability to Communicate in Primary Language [Count of Participants; unit: Participants]
  Not At All | 0 | 1 | 0 | 1
  Very Well | 3 | 17 | 19 | 39
If Participant Speaks Second Language, Ability to Very Well Communicate in Second Language [Count of Participants; unit: Participants] — Population: Analysis was performed only on participants who were able to speak second language.
  Participants
    number analyzed (Participants) | 0 | 18 | 0 | 18
    (all) | 0 | 1 | 0 | 1
Does Participant Speak More Than Two Languages [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 0 | 1
  No | 3 | 17 | 19 | 39
Diabetic Status [Count of Participants; unit: Participants]
  Diabetic | 0 | 3 | 3 | 6
  Non-Diabetic | 3 | 15 | 16 | 34
Baseline Statin Use [Count of Participants; unit: Participants]
  Yes | 1 | 9 | 8 | 18
  No | 2 | 9 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Extension Study Baseline in Composite Score of a Broad Cognitive Test Battery at Month 24
Description: Composite scores were derived from the test battery. Each test in the battery falls into 1 of the following cognitive domains: Episodic Memory (California Verbal Learning Test - 2nd Edition [CVLT-II], Brief Visuospatial Memory Test - Revised [BVMT-R]), Executive Function (Trail Making Part B, Digit Span Backwards), Language (Animals, Lexical/Phonemic Fluency), Attention (Digit Span Forward, Trail Making Part A), and Visuospatial (Clock Drawing, BVMT-Copy). Only the domains of episodic memory, executive function, language, and attention were used for the calculation of composite score (i.e., Clock Drawing, BVMT-Copy, and the Multilingual Naming Test (MINT), which do not allow generation of standard z scores, were only used for diagnostic purposes and were excluded from the calculation of the composite score). To form the composite, z-scores were calculated for each test, each z-score for the domain were averaged, and then all relevant domains were averaged to form the composite.
Time Frame: Baseline and Month 24
Population: As the study was early terminated, there were limited number of enrolled participants and insufficient treatment duration, therefore, data was not collected for this outcome measure.
Groups:
- High Risk Pioglitazone 0.8 mg: Pioglitazone 0.8 mg tablets, orally, once daily for 3 years to participants assigned to high risk group for developing MCI- AD within the next five years in previous study (AD-4833/TOMM40_301).
Arm/Group | Low Risk Placebo | High Risk Placebo | High Risk Pioglitazone 0.8 mg
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Time to Diagnosis of Alzheimer's Disease (AD) Dementia
Time Frame: Day 1 and every 6 months (up to maximum of 36 months)
Population: as for outcome 1
Arm/Group | Low Risk Placebo | High Risk Placebo | High Risk Pioglitazone 0.8 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after receiving the last dose of study drug (approximately up to 1113 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Low Risk Placebo | High Risk Placebo | High Risk Pioglitazone
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/3 | 4/18 | 3/19
Other Adverse Events (participants affected / at risk) | 1/3 | 10/18 | 12/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Risk Placebo (N=3) | High Risk Placebo (N=18) | High Risk Pioglitazone (N=19)
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Risk Placebo (N=3) | High Risk Placebo (N=18) | High Risk Pioglitazone (N=19)
Cataract (Eye disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 4
Urinary tract infection (Infections and infestations) | 0 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT02284906/SAP_000.pdf
  • Study Protocol (2016-01-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT02284906/Prot_001.pdf